CLINICAL TRIAL: NCT00180375
Title: OPERA: French Observational Study on Patients Implanted With a Guidant PRIZM or Vitality Defibrillator
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: OPERA Registry; 902194
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Ventricular Tachycardia; Ventricular Fibrillation
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation | interventions — Defibrillators, Implantable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Prizm, Vitality, Renewal — Follow-up during 2 years
  Other Names: ICD and CRT-D

SUMMARY:
This study evaluates the date of the first appropriate and/or inappropriate therapy in patients implanted with a Guidant PRIZM or VITALITY defibrillator and is evaluating eventual predictive risk factors for appropriate/inappropriate therapies as well as the influence of the programmed parameters on these therapies.

DETAILED DESCRIPTION:
The registry measured the times to, and studied the determinants of, first appropriate (FAT) and inappropriate (FIT) therapy delivered by single, dual and triple chamber (CRT-D) ICD implanted for primary and secondary prevention indications.

ELIGIBILITY:
Inclusion Criteria:

* Indication for an ICD according to current guidelines, incl. prophylactic indication

Exclusion Criteria:

* pregnant or at birth bearing age without contraception, participation in another clinical trial, short life expectancy, geographically unstable for a follow-up at the investigational center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a conventional indication of ICD or CRT-D
Sampling Method: Non-Probability Sample
Enrollment: 636 (Actual)
Dates: Start 2002-05; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Time to first appropriate therapy | 2 year-follow-up
Time to first inappropriate therapy | 2 year-follow-up

SECONDARY OUTCOMES:
Influence of cardiopathy, EF, NYHA Class, Type of ventricular arrhythmia (MVT, PVT, VF), History of atrial and ventricular arrhythmias, medical treatment (betablockers and/or Amiodarone). | 2 year-follow-up
Type of treatment ATP/shock | 2 year-follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Antoine LEENHARD, MD, Principal Investigator — Hôpital Lariboisière, Paris
Locations (33):
- France (33):
  - CHG Aix en Provence, Aix-en-Provence
  - CHG Albi, Albi
  - CH Amiens, Amiens
  - CHU Angers, Angers
  - Hopital Angouleme, Angoulême
  - CH Avignon, Avignon
  - CH Besancon, Besançon
  - CHU Hopital la Cavale Blanche, Brest
  - Hopital Cote de Nacre, Caen
  - CHG Chateauroux, Châteauroux
  - Hopital Antoine Beclere, Clamart
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CHU Michalon, Grenoble
  - CH La Roche sur Yon, La Roche-sur-Yon
  - CHU Dupuytren, Limoges
  - Hopital Neuro-cardiologique, Lyon
  - CH St. Joseph, Marseille
  - GH La Timone, Marseille
  - Hopital Nord, Marseille
  - CHG Martigues, Martigues
  - Hôpital Princesse de Grâce, Monaco
  - CHU Montpellier, Montpellier
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - CHU D'Orleans, Orléans
  - CHG Pau, Pau
  - CHRU Robert Debré, Reims
  - CHU Pontchaillou, Rennes
  - CHU Rouen, Rouen
  - CMC Arnaud Tzanck, Saint-Laurent-du-Var
  - CHU Toulon, Toulon
  - CHU Rangueil, Toulouse
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No